CLINICAL TRIAL: NCT07177469
Title: A Phase II Study to Evaluate the Efficacy and Safety of UBT251 Injection in Overweight/Obese Patients
Brief Title: UBT251 Injection Phase II Study (Overweight or Obesity)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The United Bio-Technology (Hengqin) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUL-UBT251(Ⅱ-1)202404
Record Dates: First submitted 2025-09-01; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UBT251 Injection 2.0 mg (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 0.5 mg subcutaneous injection with increasing doses at 5, 9weeks to 1.0 mg and 2.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 2.0 mg and UBT251 Injection Placebo
- UBT251 Injection 4.0 mg（ID 0.5 mg） (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 0.5 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 1.0 mg, 2.0 mg and 4.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 4.0 mg (ID 0.5 mg) and UBT251 Injection Placebo
- UBT251 Injection 4.0 mg（ID 1.0 mg） (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 1.0 mg subcutaneous injection with increasing doses at 5 and 9 weeks to 2.0 mg and 4.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 4.0 mg (ID 1.0 mg) and UBT251 Injection Placebo
- UBT251 Injection 6.0 mg (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 1.0 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 2.0 mg, 4.0 mg and 6.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 6.0 mg and UBT251 Injection Placebo

INTERVENTIONS:
Drug: UBT251 Injection 2.0 mg and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo subcutaneously once weekly
  Arms: UBT251 Injection 2.0 mg
Drug: UBT251 Injection 4.0 mg (ID 0.5 mg) and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo subcutaneously once weekly
  Arms: UBT251 Injection 4.0 mg（ID 0.5 mg）
Drug: UBT251 Injection 4.0 mg (ID 1.0 mg) and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo subcutaneously once weekly
  Arms: UBT251 Injection 4.0 mg（ID 1.0 mg）
Drug: UBT251 Injection 6.0 mg and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo subcutaneously once weekly
  Arms: UBT251 Injection 6.0 mg

SUMMARY:
This randomized, double-blind, parallel, placebo-controlled phase II study to evaluate the efficacy and safety of UBT251 Injection in overweight/obese patients

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive, of any gender;
2. Body mass index (BMI) ≥28.0 kg/m² or 24.0 kg/m² ≤ BMI < 28.0 kg/m² accompanied by at least one of the following: a. Prediabetes, hypertension, dyslipidemia, or fatty liver; b. Weight-bearing joint pain; c. Obesity-induced dyspnea or obstructive sleep apnea syndrome;
3. Stable body weight for 3 months prior to screening;
4. No fertility plans from screening to 6 months after study completion, willing to use contraceptive measures, and no sperm or egg donation plans within 6 months after study completion;
5. Fully informed about the study and voluntarily signed the written informed consent form.

Exclusion Criteria:

1. Known hypersensitivity to the investigational drug or its formulation excipients, or to other GLP-1 receptor agonist drugs, or a history of clinically significant multiple or severe drug allergies, or current allergic diseases, or high sensitivity constitution;
2. History of use of any of the following drugs or treatments within the specified periods prior to screening: 1) GLP-1 receptor agonists, GLP-1R/GCGR agonists, or GLP-1R/GIPR/GCGR agonists within 3 months before screening; 2) Over-the-counter weight-loss drugs or appetite suppressants within 3 months before screening, or prescription weight-loss drugs or lipolytic injectables within 3 months before screening; 3) Drugs likely to affect body weight (e.g.systemic glucocorticoids, tricyclic antidepressants, antipsychotics, or antiepileptics) for ≥2 consecutive weeks within 3 months before screening or expected during the trial; 4) Antidiabetic drugs (e.g.metformin, SGLT2 inhibitors,thiazolidinediones) within 3 months before screening;
3. History or evidence of any of the following diseases: 1) Diagnosis of type 1 diabetes, type 2 diabetes, or other types of diabetes; 2) History of acute or chronic pancreatitis or pancreatic surgery; 3) Symptomatic gallbladder disease within 2 years before screening (defined as imaging evidence of gallstones with doctor-diagnosed abdominal pain attributable to gallstones); subjects who have undergone cholecystectomy and/or cholelithiasis treatment without long-term complications may participate; 4) Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2; 5) Secondary obesity due to disease or medication; 6) History of bariatric surgery (excluding: acupuncture for weight loss, liposuction, or abdominal liposuction performed >1 year before screening; gastric banding removed >1 year before screening; intragastric balloon removed >1 year before screening; duodenal-jejunal bypass sleeve removed >1 year before screening); 7) History of depression or Patient Health Questionnaire-9 (PHQ-9) score ≥15 at screening; or history of severe mental illness (including suicidal ideation/attempts, schizophrenia, bipolar disorder, etc.); 8) Clinically significant cardiovascular disease within 6 months before screening (defined as: i. Myocardial infarction or unstable angina; ii. Cardiac surgery; iii. Congestive heart failure; iv. Cerebrovascular accident, including stroke/transient ischemic attack; v. Other cardiovascular diseases deemed unsuitable for the trial by the investigator); 9) History of retinal disease; 10) History of severe hypoglycemia or recurrent symptomatic hypoglycemia; 11) Concurrent gastroparesis or other gastrointestinal motility disorders, uncontrolled gastroesophageal reflux disease, or gastrointestinal diseases that increase the risk of adverse events with medication use; 12) Major surgery, severe trauma, or severe infection within 1 month before screening, as judged by the investigator to be unsuitable for the trial; 13) History of malignant tumors; 14) Limb deformities or disabilities that prevent accurate measurement of height, weight, or other indicators; 15) Concurrent diseases (e.g.neurological, endocrine, mental diseases) that, in the investigator's opinion, may affect subject safety, efficacy evaluation, or compliance;
4. Screening abnormalities in any of the following tests: 1) HbA1c ≥6.5% or fasting blood glucose (FBG) ≥7.0 mmol/L; if FBG is 6.1-6.9 mmol/L at screening, an oral glucose tolerance test (OGTT) is required, and subjects with 2-hour post-load blood glucose ≥11.1 mmol/L will be excluded; 2) Hepatic or renal impairment (serum ALT and/or AST ≥3 times the upper limit of normal [ULN]; serum total bilirubin ≥1.5×ULN; estimated glomerular filtration rate [eGFR] <60 mL·min-¹·1.73m-² according to local laboratory reference ranges); 3) Serum calcitonin ≥50 pg/mL; 4) Thyroid dysfunction (confirmed by clinical assessment and/or abnormal thyroid-stimulating hormone [TSH]) with hyperthyroidism or hypothyroidism that may increase patient risk; 5) Fasting triglycerides ≥5.6 mmol/L; 6) Serum amylase or lipase >2.0×ULN; 7) International normalized ratio (INR) above the normal range at screening; 8) Hemoglobin <110 g/L (male) or <100 g/L (female); 9) Untreated or poorly controlled hypertension; 10) Clinically significant electrocardiogram (ECG) abnormalities at screening; 11) Diagnosis of hypokalemia or hypomagnesemia at screening; 12) Physical examination, vital signs, or laboratory findings with clinically significant abnormalities that, in the investigator's judgment, pose a major risk to the subject or interfere with safety, pharmacokinetic (PK), or pharmacodynamic (PD) result evaluation;
5. Positive hepatitis B surface antigen (HBsAg) with hepatitis B virus (HBV) deoxyribonucleic acid (DNA) above the reference value, positive hepatitis C virus (HCV) antibody with HCV ribonucleic acid (RNA) exceeding the reference range upper limit, positive human immunodeficiency virus (HIV) antibody, or positive syphilis antibody at screening;
6. Blood loss or blood donation exceeding 400 mL within 3 months before screening, or receipt of blood or blood component transfusions; or concurrent hemoglobinopathies, hemolytic anemia, or sickle cell anemia;
7. Participation in other clinical trials within 3 months before screening;
8. History of drug or alcohol abuse, defined as female subjects consuming >7 standard drinks per week or male subjects consuming >14 standard drinks per week;
9. Pregnant or lactating women;
10. Inability to tolerate venipuncture or history of fainting or dizziness during blood draws;
11. Other conditions deemed unsuitable for participation in the clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Week 24
  Percentage change in body weight from baseline after 24 weeks of treatment

SECONDARY OUTCOMES:
Waist Circumference | Week 24
  change in waist circumference from baseline after 24 weeks of treatment
BMI | Week 24
  change in BMI from baseline after 24 weeks of treatment
Fasting Serum Lipids | Week 24
  change in fasting serum lipids from baseline after 24 weeks of treatment
Systolic blood pressure | Week 24
  change in systolic blood pressure from baseline after 24 weeks of treatment
Diastolic blood pressure | Week 24
  change in diastolic blood pressure from baseline after 24 weeks of treatment
HbA1c | Week 24
  change in HbA1c from baseline after 24 weeks of treatment
Adverse Events | Through study completion, an average of six months
  The incidence of Adverse Event (AE), Adverse Event of Special Interest (AESI), Adverse Drug Reaction (ADR), Serious Adverse Event (SAE) and withdrawal due to Adverse Events
Mental Health Status | Through study completion, an average of six months
  Changes in mental health status which will be evaluated using the PHQ-9 scale
Plasma Concentration | Through study completion, an average of six months
  Plasma Concentration of UBT251 at different time point
Serum Anti-UBT251 Antibody Incidence | Through study completion, an average of six months
  Change in serum anti-UBT251 antibody incidence
Titre and neutralizing antibody testing of antibody-positive samples | Through study completion, an average of six months
  change in titre and neutralizing antibody testing of antibody-positive samples
ECG | Through study completion, an average of six months
  change in components of the ECG (e.g. QRS Complex, QT Interval, etc.)
Respiration in breaths per minute by investigator | Through study completion, an average of six months
  change in respiration in breaths per minute by investigator
Temperature in degree Celsius by thermometer | Through study completion, an average of six months
  change in temperature in degree Celsius by thermometer
Pulse in beats per minute by investigator | Through study completion, an average of six months
  change in pulse in beats per minute as measured by the investigator
Abnormal findings in physical examination by investigator | Through study completion, an average of six months
  change in physical examination by investigator which includes the skin, lymph nodes, head, neck, heart, lungs, abdomen, umbilical region, and spine/limbs. Abnormal findings from the physical examination will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No